CLINICAL TRIAL: NCT04545749
Title: A Phase I, Open-label Study to Evaluate the Safety, Tolerability, and Immunogenicity of UB-612 Vaccine in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of UB-612 COVID-19 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical Inc., Asia (Industry)
Collaborators: Vaxxinity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: V-122
Record Dates: First submitted 2020-09-02; First posted 2020-09-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — UB-612 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Low dose) (Experimental): 20 subjects will be enrolled to receive low dose of UB-612 vaccine.
  Interventions: Biological: UB-612
- Group B (Medium dose) (Experimental): 20 subjects will be enrolled to receive medium dose of UB-612 vaccine.
  Interventions: Biological: UB-612
- Group C (High dose) (Experimental): 20 subjects will be enrolled to receive high dose of UB-612 vaccine.
  Interventions: Biological: UB-612

INTERVENTIONS:
Biological: UB-612 — UB-612 is a proprietary high-precision designer S1-RBD-protein based vaccine incorporating a Th/CTL epitope peptide pool which could bind to human MHC-I and MHC-II to activate T cells.

SUMMARY:
This is a phase I, open-label, dose-escalation clinical study to evaluate the safety, tolerability and immunogenicity of 3 ascending doses of UB-612 COVID-19 vaccine in healthy adults, aged from 20 to 55 years old.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation clinical study to evaluate the safety, tolerability and immunogenicity of 3 ascending doses of UB-612 COVID-19 vaccine in healthy adults. Up to 60 subjects (20 subjects per group) will be enrolled into this study. Subjects in each group will be enrolled to receive two doses of UB-612 vaccine at 28-day interval (Day 0 and Day 28).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female between the age of 20 and 55 years at time of enrollment.
2. Women of childbearing potential and men must agree to practice medically effective contraception from first vaccination until 3 months after the last vaccination.
3. Able to understand the content and possible risks of informed consent and willing to sign the Informed Consent Form (ICF).
4. Able to understand and agrees to comply with all study procedures and be available for all study visits.
5. Negative serological test for Hepatitis B surface antigen (HBsAg), HCV RNA and HIV antibody screening.
6. Negative in serum antibodies (IgG) against SARS-CoV-2 ELISA.
7. Negative result of RT-PCR screening of nasopharyngeal or throat swabs for SARS-CoV-2.
8. Ear temperature ≤ 38.0°C.
9. The body mass index (BMI) of 18-30 kg/m2, inclusive, at screening.
10. Indexes of blood routine, biochemistry and other laboratory tests are within the normal ranges, or not clinically significant as judged by investigators.
11. Judged to be healthy by the investigator on the basis of medical history, physical examination, 12-lead ECG, vital signs, and clinical laboratory tests performed at screening.

Exclusion Criteria:

1. History of anaphylaxis, urticarial, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
2. Female who is pregnant or positive in pregnancy test at screening or just prior to each vaccination administration.
3. Female who is breast-feeding or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
4. Any acute illness, as determined by the study investigator 3 days before first vaccination.
5. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
6. Known history of SARS or MERS.
7. Previous exposure to SARS-CoV-2 or receipt of an investigational vaccine product for the prevention of COVID-19, MERS or SARS.
8. Subjects who take part in another clinical study within 12 weeks prior to the day of informed consent.
9. With certain underlying medical conditions which are at increased risk for severe illness from COVID-19.
10. Congenital or acquired angioedema.
11. Immune deficiency/disorder, whether due to genetic defect, immunodeficiency disease or immunosuppressive therapy.
12. Platelet disorder or other bleeding disorder may cause injection contraindication.
13. Prior chronic administration of immunosuppressant or corticosteroids, cytotoxic treatment in last 6 months before first vaccination.
14. Prior administration of immunoglobulins and/or any blood products in last 4 months before first vaccination.
15. Prior administration of attenuated, nucleic acid (mRNA or DNA) or vectored vaccines in last 1 month before first vaccination or expectation of such vaccines in the month after the second vaccination.
16. Prior administration of subunit vaccine or inactivated vaccine in last 14 days before first vaccination or expectation of receipt of such vaccines in the 14 days after the second vaccination.
17. Current anti-tuberculosis (TB) therapy or history of TB.
18. Alcoholism or substance abuser.
19. History of malignancy within 5 years prior to screening visit, except basal cell carcinoma of the skin and cervical carcinoma in situ.
20. Any medical disease or condition that, in the opinion of the study investigator, may confound the results of the study or pose an additional risk to the subjects by their participation in the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Safety of UB-612 vaccine | 7 days following vaccination
  1. Occurrence of adverse reactions within 7 days after vaccination
  2. Percentage of subjects with ≥ Grade 3 adverse events within 7 days after vaccination

SECONDARY OUTCOMES:
Safety | Day 0 to Day 56
  1. Occurrence of adverse events (AEs) till Day 56
  2. Occurrence of serious adverse events (SAEs) till Day 56
Safety | Day 29 to Day 196
  Occurrence of serious adverse events during the whole follow-up period
Safety | Day 0 to Day 196
  Occurrence of adverse events of special interest during the study period
Immunogenicity | Day 14, 28, 42, 56, 112, and 196
  Geometric mean titer (GMT) of antigen-specific antibody (Anti-S1-RBD)
Immunogenicity | Day 14, 28, 42, 56, 112, and 196
  Seroconversion rate (SCR) of antigen-specific antibody (Anti-S1-RBD)
Immunogenicity | Day 14, 28, 42, 56, 112, and 196
  Geometric mean fold increase of antigen-specific antibody (Anti-S1-RBD)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Yi Wang, Ph.D., Study Chair — United Biomedical Inc., Asia
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Wang CY, Hwang KP, Kuo HK, Peng WJ, Shen YH, Kuo BS, Huang JH, Liu H, Ho YH, Lin F, Ding S, Liu Z, Wu HT, Huang CT, Lee YJ, Liu MC, Yang YC, Lu PL, Tsai HC, Lee CH, Shi ZY, Liu CE, Liao CH, Chang FY, Chen HC, Wang FD, Hou KL, Cheng J, Wang MS, Yang YT, Chiu HC, Jiang MH, Shih HY, Shen HY, Chang PY, Lan YR, Chen CT, Lin YL, Liang JJ, Liao CC, Chou YC, Morris MK, Hanson CV, Guirakhoo F, Hellerstein M, Yu HJ, King CC, Kemp T, Heppner DG, Monath TP. A multitope SARS-CoV-2 vaccine provides long-lasting B cell and T cell immunity against Delta and Omicron variants. J Clin Invest. 2022 May 16;132(10):e157707. doi: 10.1172/JCI157707. PMID 35316221